CLINICAL TRIAL: NCT03198715
Title: A Phase I, Single Blind, Placebo-controlled, Randomized Study to Assess the Safety of DS-1040b in Subjects With Thrombectomy Treated Acute Ischemic Stroke.
Brief Title: Safety of DS-1040b in Acute Ischemic Stroke Patients Treated With Thrombectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: DS1040-A-J110; 173612 (Registry Identifier: JAPIC CTI)
Record Dates: First submitted 2017-06-19; First posted 2017-06-26 (Actual); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Fibrinolysis enhancer; TAFIa inhibitor; Developmental Phase I
MeSH Terms: conditions — Ischemic Stroke | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- DS-1040b 0.6 mg (Experimental): Participants receive DS-1040b 0.6 mg by intravenous infusion over six hours
  Interventions: Drug: DS1040b
- DS-1040b 1.2 mg (Experimental): Participants receive DS-1040b 1.2 mg by intravenous infusion over six hours
  Interventions: Drug: DS1040b
- DS-1040b 2.4 mg (Experimental): Participants receive DS-1040b 2.4 mg by intravenous infusion over six hours
  Interventions: Drug: DS1040b
- DS-1040b 4.8 mg (Experimental): Participants receive DS-1040b 4.8 mg by intravenous infusion over six hours
  Interventions: Drug: DS1040b
- Placebo (Placebo Comparator): Participants receive saline by intravenous infusion over six hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DS1040b — DS-1040b in solution for intravenous infusion
  Other Names: Investigational product
  Arms: DS-1040b 0.6 mg; DS-1040b 1.2 mg; DS-1040b 2.4 mg; DS-1040b 4.8 mg
Drug: Placebo — Saline solution for intravenous infusion
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
The aim of this study is to find out if DS-1040b is safe and tolerable in acute ischemic stroke patients with thrombectomy. Four groups will receive different doses of DS-1040b by intravenous infusion for 6 hours. Groups with the lowest dose will start. When it is determined that each dose is safe and tolerable, the next higher dose will be given to the next group.

ELIGIBILITY:
Inclusion Criteria:

* Is an acute ischemic stroke patients with evidence of intracranial vascular occlusion
* Is enrolled in principle within 8 hours of symptom onset
* Has treatment plan that includes stent retriever
* Has protocol-defined scores on several scales

Exclusion Criteria:

* Has treatment plan that includes fibrinolysis or fibinolysis
* Has identified intracranial hemorrhage or subarachnoid hemorrhage
* Has active bleeding like gastrointestinal hemorrhage
* Has cerebral bleeding risk; intracranial tumor, brain aneurysm, cerebral arteriovenous malformation, or history of intracranial bleeding
* Has severe hepatic or renal impairment
* Has been a participant in other clinical trial within 30 days prior to treatment
* Is pregnant, lactating, or planning on becoming pregnant during treatment period
* Has any condition or history that might, per protocol or in the opinion of the investigator, compromise:

  1. safety or well-being of the participant or their offspring
  2. safety of the study staff
  3. analysis of results

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-07-30 (Actual); Primary Completion 2020-01-19 (Actual); Study Completion 2020-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (20):
- Japan (20):
  - Hirosaki University Hospital, Hirosaki, Aomori
  - Funabashi Municipal Medical Center, Funabashi, Chiba
  - Kokura Memorial Hospital, Kitakyushu, Fukuota
  - Mihara Memorial Hospital, Isesaki, Gunma
  - Nakamura Memorial Hospital, Sapporo, Hokkaido
  - Japan Organization of Occupational Health and Safety Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Hyogo College of Medicine College Hospital, Nishinomiya, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Iwate Prefectural Central Hospital, Morioka, Iwate
  - Seisho Hospital, Odawara, Kanagawa
  - Yokohama Municipal Citizen's Hospital, Yokohama, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Nagasaki University Hospital, Nagasaki
  - Niigata City General Hospital, Niigata
  - Wakayama Medical University Hospital, Wakayama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sakai N, Takeuchi M, Imamura H, Shimamura N, Yoshimura S, Naito H, Kimura N, Masuo O, Hirotsune N, Morita K, Toyoda K, Yamagami H, Ishihara H, Nakatsu T, Miyoshi N, Suda M, Fujimoto S. Safety, Pharmacokinetics and Pharmacodynamics of DS-1040, in Combination with Thrombectomy, in Japanese Patients with Acute Ischemic Stroke. Clin Drug Investig. 2022 Feb;42(2):137-149. doi: 10.1007/s40261-021-01112-8. Epub 2022 Jan 21. PMID 35061236

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 42 participants who met all inclusion criteria and no exclusion criteria were randomized to treatment. Of the 42 participants randomized, 41 participants received treatment.
Pre-assignment Details: The study consisted of 4 parallel, ascending-dose cohorts. The DS-1040b 0.6 mg cohort only consisted of a DS-1040b group. A ratio of DS-1040b:placebo of 3:1 per cohort was used for the 1.2 mg and higher dose cohorts.
Groups:
- DS-1040b 0.6 mg: Participants who received a single, intravenous infusion of DS-1040b 0.6 mg.
- DS-1040b 1.2 mg: Participants who received a single, intravenous infusion of DS-1040b 1.2 mg.
- DS-1040b 2.4 mg: Participants who received a single, intravenous infusion of DS-1040b 2.4 mg.
- DS-1040b 4.8 mg: Participants who received a single, intravenous infusion of DS-1040b 4.8 mg.
- Placebo: Participants who received a single, intravenous infusion of placebo.
Period: Overall Study
Arm/Group | DS-1040b 0.6 mg | DS-1040b 1.2 mg | DS-1040b 2.4 mg | DS-1040b 4.8 mg | Placebo
Started | 6 | 12 | 12 | 3 | 9
Completed | 6 | 11 | 10 | 3 | 7
Not Completed | 0 | 1 | 2 | 0 | 2
Not completed — Death | 0 | 0 | 1 | 0 | 2
Not completed — Other | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographics and baseline characteristics were assessed in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | DS-1040b 0.6 mg | DS-1040b 1.2 mg | DS-1040b 2.4 mg | DS-1040b 4.8 mg | Placebo | Total
Number analyzed (Participants) | 6 | 12 | 11 | 3 | 9 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2 | 1 | 1 | 6
  >=65 years | 5 | 11 | 9 | 2 | 8 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (6.80) | 76.3 (6.96) | 73.6 (10.40) | 69.0 (7.81) | 76.9 (11.22) | 74.5 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 5 | 2 | 5 | 19
  Male | 4 | 7 | 6 | 1 | 4 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 12 | 11 | 3 | 9 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 12 | 11 | 3 | 9 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 6 | 12 | 11 | 3 | 9 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Symptomatic or Asymptomatic Intracranial Hemorrhage (ICH) Within 36 Hours From Start of Treatment With DS-1040b in Acute Ischemic Stroke Participants
Description: Symptomatic and asymptomatic intracranial hemorrhage (ICH) confirmed by head imaging (CT or MRI) are reported. Symptomatic ICH was defined as Intracranial hemorrhage with clinical deterioration causing an increase in the National Institutes of Health Stroke Scale (NIHSS) score of ≥ 4 points (defined by European Cooperative Acute Stroke Study). Asymptomatic ICH included the following: Hemorrhagic infarction type 1: Small petechial hemorrhage along the margins of the infarct, Hemorrhagic infarction type 2: Confluent petechial hemorrhage within the infarcted area, but without a mass effect, Parenchymal hematoma type 1: Hematoma involving ≤ 30% of the infarcted area with a slight mass effect, Parenchymal hematoma type 2: Hematoma involving > 30% of, or outside the infarcted area, with a significant mass effect.
Time Frame: From start of treatment up to 36 hours post single, intravenous dose
Population: Bleeding events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-1040b 0.6 mg | DS-1040b 1.2 mg | DS-1040b 2.4 mg | DS-1040b 4.8 mg | Placebo
Number analyzed (Participants) | 6 | 12 | 11 | 3 | 9
Participants
  Symptomatic ICH | 0 | 0 | 0 | 0 | 0
  Asymptomatic ICH | 2 | 5 | 4 | 1 | 1
  Hemorrhagic infarction type 1 | 0 | 1 | 0 | 0 | 0
  Hemorrhagic infarction type 2 | 1 | 1 | 1 | 0 | 0
  Parenchymal hematoma type 1 | 0 | 3 | 0 | 1 | 0
  Parenchymal hematoma type 2 | 0 | 0 | 2 | 0 | 0
  Not applicable | 1 | 1 | 1 | 0 | 1

2. Primary Outcome: Number of Participants With Non-ICH Major Bleeding Within 96 Hours From Start of Treatment With DS-1040b In Acute Ischemic Stroke Participants
Description: Non-ICH was defined as a clinically evident bleeding with a 5 g/dL or greater decrease in hemoglobin.
Time Frame: From start of treatment up to 96 hours post single, intravenous dose
Population: Bleeding events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-1040b 0.6 mg | DS-1040b 1.2 mg | DS-1040b 2.4 mg | DS-1040b 4.8 mg | Placebo
Number analyzed (Participants) | 6 | 12 | 11 | 3 | 9
Participants | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Pharmacokinetic Analysis Area Under The Plasma Concentration Time Curve (AUC) of DS-1040a in Plasma
Description: The pharmacokinetic (PK) parameter of area under the plasma concentration-time curve up to the last quantifiable time was calculated using linear up logarithmic down rule.
Time Frame: Predose, 0.5 hours (h), 3 h, 6 h, 18 h, 24 h, 48 h, and 96 h post single, intravenous dose
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | DS-1040b 0.6 mg | DS-1040b 1.2 mg | DS-1040b 2.4 mg | DS-1040b 4.8 mg
Number analyzed (Participants) | 6 | 11 | 10 | 3
ng*h/mL | 111 (45.5) | 275 (72.2) | 570 (230) | 1550 (962)

4. Secondary Outcome: Pharmacokinetic Analysis Maximum Concentration (Cmax) of DS-1040a in Plasma
Description: The PK parameter of maximum concentration (Cmax) was observed values.
Time Frame: Predose, 0.5 hours (h), 3 h, 6 h, 18 h, 24 h, 48 h, and 96 h post single, intravenous dose
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DS-1040b 0.6 mg | DS-1040b 1.2 mg | DS-1040b 2.4 mg | DS-1040b 4.8 mg
Number analyzed (Participants) | 6 | 11 | 10 | 3
ng/mL | 17.2 (6.25) | 29.7 (7.50) | 60.6 (11.8) | 141 (61.7)

5. Secondary Outcome: Pharmacokinetic Analysis Time to Maximum Concentration (Tmax) of DS-1040b in Plasma
Description: The PK parameter of time to maximum concentration (Tmax) was observed values. When there are more than one time point, the time point when the concentration reached the first Cmax will be used as Tmax.
Time Frame: Predose, 0.5 hours (h), 3 h, 6 h, 18 h, 24 h, 48 h, and 96 h post single, intravenous dose
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | DS-1040b 0.6 mg | DS-1040b 1.2 mg | DS-1040b 2.4 mg | DS-1040b 4.8 mg
Number analyzed (Participants) | 6 | 11 | 10 | 3
hours | 2.21 (2.18) | 4.67 (2.29) | 5.11 (1.85) | 5.96 (0.03)

6. Secondary Outcome: Pharmacokinetic Analysis Terminal Half-Life (T1/2) of DS-1040b in Plasma
Description: The PK parameter of terminal half-life (T1/2) was calculated from the following formula in participants whose Kel could be calculated. T1/2=ln2 / Kel
Time Frame: Predose, 0.5 hours (h), 3 h, 6 h, 18 h, 24 h, 48 h, and 96 h post single, intravenous dose
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis set in participants with available sample for analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | DS-1040b 0.6 mg | DS-1040b 1.2 mg | DS-1040b 2.4 mg | DS-1040b 4.8 mg
Number analyzed (Participants) | 1 | 3 | 5 | 3
hours | 4.61 | 16.8 (1.74) | 19.5 (10.5) | 29.7 (2.35)

7. Secondary Outcome: Pharmacokinetic Analysis Mean Amount of DS-1040a Excreted in Urine in Acute Ischemic Stroke Participants
Description: The pharmacokinetic parameter of amount of drug excreted in urine was calculated from the following formula:
  urine concentration (ng/mL) /10^6× (urine weight / urinary specific gravity)
Time Frame: From start of treatment up to 24 hours post single, intravenous dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | DS-1040b 0.6 mg | DS-1040b 1.2 mg | DS-1040b 2.4 mg | DS-1040b 4.8 mg
Number analyzed (Participants) | 6 | 9 | 10 | 3
mg | 0.420 (0.0308) | 0.880 (0.0683) | 1.49 (0.309) | 3.45 (0.417)

8. Secondary Outcome: Pharmacodynamic Analysis Thrombin Activatable Fibrinolysis Inhibitor (TAFI) Antigen Levels in Plasma and Change From Baseline in Acute Ischemic Stroke Participants
Description: The mean thrombin activatable fibrinolysis (TAFI) antigen levels and change from baseline in TAFI levels are reported. Change from baseline is based on the number of participants with baseline and at least one post-baseline laboratory test.
Time Frame: Baseline, 6 hours and 24 hours post single, intravenous dose
Population: Pharmacodynamic parameters were assessed in the Pharmacodynamic Analysis Set.
Measure: Mean (Standard Deviation); unit: % of normal pooled plasma control
Arm/Group | DS-1040b 0.6 mg | DS-1040b 1.2 mg | DS-1040b 2.4 mg | DS-1040b 4.8 mg | Placebo
Number analyzed (Participants) | 6 | 11 | 10 | 3 | 8
% of normal pooled plasma control
  Baseline: number analyzed (Participants) | 6 | 11 | 7 | 3 | 8
  Baseline | 99.17 (25.527) | 80.05 (9.101) | 79.56 (19.553) | 81.90 (2.750) | 88.28 (17.157)
  6 hours postdose: number analyzed (Participants) | 6 | 10 | 9 | 3 | 8
  6 hours postdose | 94.05 (22.090) | 81.37 (11.358) | 86.12 (13.727) | 81.23 (6.313) | 87.55 (15.987)
  24 hours postdose | 87.75 (20.938) | 78.09 (11.033) | 77.62 (14.208) | 72.70 (8.681) | 79.11 (13.051)
  Change from baseline to 6 hour postdose: number analyzed (Participants) | 6 | 10 | 6 | 3 | 8
  Change from baseline to 6 hour postdose | -5.12 (6.463) | 1.69 (5.077) | 1.28 (8.551) | -0.67 (4.202) | -0.73 (5.579)
  Change from baseline to 24 hours postdose: number analyzed (Participants) | 6 | 11 | 7 | 3 | 8
  Change from baseline to 24 hours postdose | -11.42 (6.934) | -1.95 (9.641) | -5.09 (6.625) | -9.20 (6.070) | -9.16 (9.759)

9. Secondary Outcome: Pharmacodynamic Analysis D-dimer Levels in Plasma and Change From Baseline in Acute Ischemic Stroke Participants
Description: Mean D-dimer levels and change from baseline in D-dimer levels are reported.Change from baseline is based on the number of subjects with baseline and at least one post-baseline laboratory test.
Time Frame: Baseline, 6 hours, 24 hours, and 48 hours post single, intravenous dose
Population: Pharmacodynamic parameters were assessed in the Pharmacodynamic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug/mL FEU
Arm/Group | DS-1040b 0.6 mg | DS-1040b 1.2 mg | DS-1040b 2.4 mg | DS-1040b 4.8 mg | Placebo
Number analyzed (Participants) | 6 | 11 | 10 | 3 | 8
ug/mL FEU
  Baseline: number analyzed (Participants) | 6 | 11 | 7 | 3 | 8
  Baseline | 1.600 (2.8865) | 0.730 (0.4176) | 2.423 (4.8964) | 0.613 (0.1250) | 3.096 (6.8343)
  6 hours postdose: number analyzed (Participants) | 5 | 10 | 9 | 3 | 7
  6 hours postdose | 1.368 (2.1428) | 0.717 (0.4899) | 3.254 (6.3573) | 1.090 (0.4540) | 3.436 (7.3095)
  24 hours postdose: number analyzed (Participants) | 6 | 10 | 10 | 3 | 7
  24 hours postdose | 1.158 (1.6216) | 0.960 (0.7254) | 2.879 (6.0571) | 1.067 (0.5235) | 3.731 (7.1964)
  48 hours postdose: number analyzed (Participants) | 6 | 9 | 10 | 3 | 7
  48 hours postdose | 0.907 (1.1908) | 0.912 (0.5107) | 2.668 (6.0954) | 1.287 (0.7371) | 0.941 (0.5545)
  Change from baseline to 6 hour postdose: number analyzed (Participants) | 5 | 10 | 6 | 3 | 7
  Change from baseline to 6 hour postdose | -0.452 (1.0327) | -0.008 (0.1091) | 1.497 (2.6031) | 0.477 (0.5742) | -0.023 (0.1340)
  Change from baseline to 24 hours postdose: number analyzed (Participants) | 6 | 10 | 7 | 3 | 7
  Change from baseline to 24 hours postdose | -0.442 (1.2701) | 0.217 (0.5241) | 1.180 (2.4023) | 0.453 (0.6422) | 0.284 (0.4342)
  Change from baseline to 48 hours postdose: number analyzed (Participants) | 6 | 9 | 7 | 3 | 7
  Change from baseline to 48 hours postdose | -0.693 (1.6989) | 0.163 (0.2431) | 1.033 (2.4047) | 0.673 (0.8559) | 0.260 (0.4700)

10. Secondary Outcome: Pharmacodynamic Analysis Activated Form of Thrombin-Activatable Fibrinolysis Inhibitor (TAFIa) Activity and Change From Baseline in Acute Ischemic Stroke Participants
Description: Mean activated form of thrombin-activatable fibrinolysis inhibitor (TAFIa) and change from baseline in TAFIa are reported. Change from baseline is based on the number of subjects with baseline and at least one post-baseline laboratory test.
Time Frame: Baseline, 6 hours, 24 hours, and 48 hours post single, intravenous dose
Population: Pharmacodynamic parameters were assessed in the Pharmacodynamic Analysis Set.
Measure: Mean (Standard Deviation); unit: % of normal pooled plasma control
Arm/Group | DS-1040b 0.6 mg | DS-1040b 1.2 mg | DS-1040b 2.4 mg | DS-1040b 4.8 mg | Placebo
Number analyzed (Participants) | 6 | 11 | 10 | 3 | 8
% of normal pooled plasma control
  Baseline: number analyzed (Participants) | 6 | 11 | 7 | 3 | 7
  Baseline | 104.5 (30.68) | 81.8 (17.67) | 93.9 (28.92) | 99.0 (8.54) | 88.7 (18.99)
  6 hours postdose: number analyzed (Participants) | 5 | 10 | 10 | 3 | 8
  6 hours postdose | 110.4 (28.10) | 77.9 (18.52) | 82.7 (16.49) | 68.7 (10.97) | 95.5 (21.63)
  24 hours postdose: number analyzed (Participants) | 5 | 10 | 10 | 3 | 8
  24 hours postdose | 93.4 (29.03) | 78.7 (14.58) | 90.7 (18.67) | 91.7 (7.51) | 88.0 (16.00)
  48 hours postdose: number analyzed (Participants) | 6 | 9 | 10 | 3 | 7
  48 hours postdose | 91.2 (27.01) | 70.0 (7.09) | 84.7 (17.50) | 88.7 (6.66) | 87.6 (13.96)
  Change from baseline to 6 hours postdose: number analyzed (Participants) | 5 | 10 | 7 | 3 | 7
  Change from baseline to 6 hours postdose | -1.4 (11.04) | -2.6 (11.82) | -14.6 (16.00) | -30.3 (13.01) | 8.0 (13.24)
  Change from baseline to 24 hours postdose: number analyzed (Participants) | 5 | 10 | 7 | 3 | 7
  Change from baseline to 24 hours postdose | -6.2 (7.56) | -5.5 (15.17) | -6.4 (12.03) | -7.3 (16.04) | 0.6 (8.00)
  Change from baseline to 48 hours postdose: number analyzed (Participants) | 6 | 9 | 7 | 3 | 7
  Change from baseline to 48 hours postdose | -13.3 (9.99) | -6.9 (11.46) | -11.0 (10.92) | -10.3 (13.61) | -1.1 (13.95)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse event (TEAE) data were collected from start of treatment up to 30 days after last study dose, up to approximately 2 years 6 months.
Description: A TEAE is defined as an adverse event (AE) that is not present prior to the study and occurs after the start of study drug administration but before Day 30, or an AE that worsens in severity after the start of study drug administration but before Day 30.
Arm/Group | DS-1040b 0.6 mg | DS-1040b 1.2 mg | DS-1040b 2.4 mg | DS-1040b 4.8 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/12 | 1/11 | 0/3 | 2/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/12 | 2/11 | 0/3 | 1/9
Other Adverse Events (participants affected / at risk) | 5/6 | 10/12 | 10/11 | 2/3 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS-1040b 0.6 mg (N=6) | DS-1040b 1.2 mg (N=12) | DS-1040b 2.4 mg (N=11) | DS-1040b 4.8 mg (N=3) | Placebo (N=9)
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS-1040b 0.6 mg (N=6) | DS-1040b 1.2 mg (N=12) | DS-1040b 2.4 mg (N=11) | DS-1040b 4.8 mg (N=3) | Placebo (N=9)
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Periodontis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Respiratory moniliasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 1 | 1 | 0 | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1 | 1 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebral artery embolism (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Neurological symptom (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Parkinsonism (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhagic infarction (Vascular disorders) | 1 | 5 | 2 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 2 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Internal haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 3 | 1 | 3
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Acetonaemic vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Lip haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1 | 2 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 2 | 0 | 1
Vessel puncture site haematoma (General disorders) | 1 | 1 | 0 | 0 | 0
Puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 1
Vessel puncture site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0 | 0
ECG signs of myocardial ischaemia (Investigations) | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 2
Pharyngeal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Urethral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Urinary tract injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT03198715/Prot_SAP_000.pdf